CLINICAL TRIAL: NCT05154708
Title: Impact on the Quality of Life of Dialysis Patients of the Routine Collection of Symptoms by the Patients Themselves, with Feedback to the Dialysis Team - Pilot Study
Brief Title: Impact of the Routine Collection of Symptoms on Quality of Life in Dialysis Patients
Acronym: FSWIFT-PILOT
Status: Terminated | Type: Observational
Why Stopped: Patient recruitment for the second phase of the pilot study was too late. There is enough information to meet the study objectives.
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Agence de La Biomédecine (Other Government); Association France REIN (Unknown)
Responsible Party: Principal Investigator, Carole AYAV, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2021-A00776-35
Record Dates: First submitted 2021-11-15; First posted 2021-12-13 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Patients Reported Outcomes
Keywords: symptoms; Patients reported outcomes; dialysis patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patient Group - Phase 1: 15 to 30 patients are expected in Phase 1 for the identification of needs and expectations in relation to a systematic electronic assessment of symptoms by the patients themselves
- Health Professionals Group - Phase 1: 15 to 30 healthcare professionals are expected to participate in Phase 1 regarding the identification of needs and expectations in relation to a systematic electronic assessment of symptoms by the patients themselves
- Patient Group - Phase 2: 50 à 60 patients were expected to test a systematic electronic assessment

SUMMARY:
Chronic kidney disease (CKD) affects 85,000 people in France. Medical care for this disease represents 2% of the Health Insurance budget.

Patients on dialysis frequently experience severe or overwhelming symptoms which contributes to poor health related quality of life (HRQoL). However, taking into account the measurement of the patients' symptoms by the patients themselves would allow to improve their HRQoL by putting more emphasis on the results that matter the most to the patients. It would also improve information and decision-making between nephrology care team and patients.

Systematic use of patients reported outcomes measures (PROMs) is not widely used due to a number of barriers including logistics and feasibility.

How will the F-SWIFT Pilot project address the barriers associated with PROMs? By choosing short questionnaires to complete By providing feedback on the severity of symptoms to the dialysis team and to patients By making links to good practice recommendations included in the feedback Allowing electronic collection of PROMs The research question therefore asks whether regular symptom monitoring with feedback to dialysis staff improves dialysis patient's outcomes? To do this, a pilot study must be carried out with the following main objectives Test the feasibility of integrating electronic measurements of PROMs with feedback to the dialysis team.

Three centers are participating in this pilot study:

* The nephrology department of the Nancy CHRU
* The Lorraine Association for the Treatment of Renal Insufficiency (ALTIR)
* The nephrology department of the Nîmes University Hospital

The project will take place in 2 phases :

Phase 1 To identify the needs and expectations of patients and health professionals in relation to a systematic electronic measurement of symptoms made by the patients themselves.

Focus groups (interviews) will be conducted with patients (n=15) and healthcare professionals (n=15).

Phase 2 (n=50-60 patients) To develop and test an electronic PROMs system allowing

* Collect patients' symptoms
* Identify patients with severe symptoms
* Alert the dialysis team in case of severe symptoms
* Suggest appropriate management strategies

DETAILED DESCRIPTION:
Patients reported outcomes (PROs) are defined as any measure of a patient's health status reported directly by the patient, without interpretation by health care professionals or others. It is how the patient feels about their health condition or treatment. Although assessing patients' well-being and managing their symptoms are the foundations of clinical care, the care patients receive often does not meet their needs. For example, healthcare professionals are often unaware of the presence and severity of their patients' symptoms. The integration of PROs into clinical trials, clinical care, and quality of care assessment stems from the need to place greater emphasis on the outcomes that matter most to patients.

To date, primary clinical trial endpoints and efficacy metrics in nephrology have been dominated by objective biochemical and process measures (percentage of patients with arteriovenous fistula). These measures fail to reflect what constitutes a good outcome from the patient's perspective, and ultimately there is often very little information about how treatments or any other interventions affect the patient's experience A growing number of studies report a high frequency of symptoms in adult dialysis patients. Patients frequently present with signs of severe pain, fatigue, nausea, cramping, itching, sleep disturbance, and depression, which are strongly associated with poor quality of life. More than half of patients experience fatigue, pruritus (relentless itching), and constipation despite available effective treatments.

In nephrology, studies have focused on survival or biomarker studies and very little on interventions to improve what was a priority for patients, i.e., treating their symptoms and improving their quality of life.

Numerous experiments have been conducted in other fields such as oncology. These studies have shown a real benefit of taking into account measures of perceived health on improving symptom management, treatment side effects and patient survival. Patients for whom regular perceived health follow-up with feedback to oncologists is implemented have a better survival than with traditional follow-up. This is mainly explained by earlier identification and management of symptoms (preventing or reducing the occurrence of downstream adverse events) or side effects of chemotherapy (allowing better tolerance and adherence to the full chemotherapy regimen).

Patients with end-stage renal disease (ESRD) treated with dialysis have poorer survival than patients with certain cancers and a particularly degraded quality of life. Symptoms reported by dialysis patients are often underestimated or even unrecognized by the dialysis team for a variety of reasons. Therefore, it seems possible to improve patient management, outcome, and quality of life through better consideration of symptoms provided the dialysis team is aware of them.

Many questions are still open. Which PRO to measure? How should it be measured? How to store and use the data? How to interpret the results? How can they be integrated with other measures in patient management and treatment decisions? The impact of routine PRO measurements is controversial, especially because of methodological biases in the various studies.

A clinical trial will be set up and nested in the national RIEN registry, entitled F-SWIFT (French-Symptom monitoring WIth Feedback Trial) to improve symptom management in order to address the unmet needs of dialysis CKD patients and improve their quality of life.

The research question posed is whether regular self-reported symptom monitoring with immediate feedback and management recommendations to the dialysis team improves the outcome of dialysis patients.

The F-SWIFT study is the French side of the Australian SWIFT study which has obtained funding and started in 2019.

irst, some technical and logistical feasibility questions need to be answered to adapt the SWIFT study to the French context. Indeed, to date, the PRO measurement is not a routine measurement in dialysis facilities. It therefore seems important to approach patients and professionals to explore their expectations and needs in terms of integrating PRO as a routine management indicator. The first phase is therefore the realization of a pilot study, which is the subject of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* For the focus group phase:

Patients

* Adult patients (≥ 18 years of age), volunteers with end-stage renal disease (ESRD) treated by dialysis in the study centers
* Individuals who have received complete information on the organization of the research and who have not objected to their participation and to the use of their data
* Person with internet access and a computer tool such as a tablet, computer or smartphone

Health professionals - Volunteer healthcare professionals in the participating departments (CHRU Nancy, ALTIR, CHU Nîmes) with at least 3 months experience in a dialysis department

For the test phase of symptom collection in dialysis services:

* Adult patients (≥ 18 years of age), volunteers with end-stage chronic kidney disease (ESRD) treated with dialysis for at least 3 months in the study participating centers
* Person who has received full information on the organization of the research and has not objected to his or her participation and to the use of his or her data
* Patient able to answer a self-questionnaire
* Person with internet access and a computer tool such as a tablet, computer or smartphone
* Person able to use a computer tool such as a tablet or smartphone
* Person affiliated to a social security system

Exclusion Criteria:

The non-inclusion criteria for the focus group phase are as follows :

Patients

* Non-dialysis patient
* Dialysis patient in retreat at the facility
* Patient dialyzed for less than 3 months
* Non-voluntary patient
* Minor patient
* Patient who does not speak French
* Person placed under judicial protection, guardianship or curatorship

Health Professionals

- Non-voluntary health professional

The non-inclusion criteria for the test phase of the collection are as follows:

* Non-dialysis patient
* Dialysis patient in retreat at the facility
* Patient dialyzed for less than 3 months
* Non-voluntary patient
* Minor patient
* Person placed under court protection, guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * For the first part
  * Patients of both sexes, of different ages and treated by dialysis (hemodialysis and peritoneal dialysis) in different structures (heavy center, medicalized dialysis unit, self-dialysis, home).
  * Health professionals: nephrologist, health executive, dialysis nurse and nurse coordinator (IPA advanced practice nurse), nursing assistants.
  * For the second part
  * Adult patients, volunteers and dialyzed in one of the participating centers: the two heavy centers of the CHRU of Nancy and Nîmes and the off-center dialysis units of ALTIR,
  * For the pilot phase, we plan to include between 50 and 60 patients (10 per heavy center, 15 in MDU, 15 in AD and 15 at home)
  Translated with www.DeepL.com/Translator (free version)
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
The feasibility of integrating electronic measurements of self-perceived symptoms with feedback to the dialysis team. | 11 months
  Feasability will be assessed through interviews with patients and health professionals. These interviews will help to identify the elements (interest in the measurement of symptoms by the patients themselves, type of symptoms to be collected, time of measurement, frequency of repetition of the measurement, alert threshold, management of alerts, management of reminders, recommendations for management, etc.) that will guarantee good acceptability of the integration of these measures.
  The feasibility will be apprehended by a test phase of the measurement of the symptoms perceived by the patients in real situation using a questionnaire given to the patients and the health professionals.

SECONDARY OUTCOMES:
Results of the focus groups with patients and health professionals | 2 months
  Identify the needs and expectations of patients and health care professionals with respect to a systematic electronic assessment of symptoms by patients themselves
Creation of the electronic symptom collection tool, implementation of links with the REIN registry, systems for managing reminders, alerts, reporting and referrals to management recommendations | 6 months
  Develop the IT tool and interface allowing :
  * the link with DIADEM* (secure connection, identity vigilance, integration of the perceived health measure in the registry),
  * the collection of symptoms,
  * identification of patients with severe symptoms,
  * alerting the dialysis team in case of severe symptoms,
  * the concomitant proposal of adapted management strategies

CONTACTS AND LOCATIONS:
Overall Officials: Luc FRIMAT, Principal Investigator — CHRU de Nancy; Olivier Moranne, Principal Investigator — Centre Hospitalier Universitaire de Nīmes; Nelly CASTIN, Principal Investigator — ALTIR
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] U.S. Department of Health and Human Services FDA Center for Drug Evaluation and Research; U.S. Department of Health and Human Services FDA Center for Biologics Evaluation and Research; U.S. Department of Health and Human Services FDA Center for Devices and Radiological Health. Guidance for industry: patient-reported outcome measures: use in medical product development to support labeling claims: draft guidance. Health Qual Life Outcomes. 2006 Oct 11;4:79. doi: 10.1186/1477-7525-4-79. PMID 17034633
- [Background] Evangelidis N, Tong A, Manns B, Hemmelgarn B, Wheeler DC, Tugwell P, Crowe S, Harris T, Van Biesen W, Winkelmayer WC, Sautenet B, O'Donoghue D, Tam-Tham H, Youssouf S, Mandayam S, Ju A, Hawley C, Pollock C, Harris DC, Johnson DW, Rifkin DE, Tentori F, Agar J, Polkinghorne KR, Gallagher M, Kerr PG, McDonald SP, Howard K, Howell M, Craig JC; Standardized Outcomes in Nephrology-Hemodialysis (SONG-HD) Initiative. Developing a Set of Core Outcomes for Trials in Hemodialysis: An International Delphi Survey. Am J Kidney Dis. 2017 Oct;70(4):464-475. doi: 10.1053/j.ajkd.2016.11.029. Epub 2017 Feb 24. PMID 28238554
- [Background] Sautenet B, Tong A, Williams G, Hemmelgarn BR, Manns B, Wheeler DC, Tugwell P, van Biesen W, Winkelmayer WC, Crowe S, Harris T, Evangelidis N, Hawley CM, Pollock C, Johnson DW, Polkinghorne KR, Howard K, Gallagher MP, Kerr PG, McDonald SP, Ju A, Craig JC. Scope and Consistency of Outcomes Reported in Randomized Trials Conducted in Adults Receiving Hemodialysis: A Systematic Review. Am J Kidney Dis. 2018 Jul;72(1):62-74. doi: 10.1053/j.ajkd.2017.11.010. Epub 2018 Feb 21. PMID 29475768
- [Background] Davison SN, Jhangri GS. Impact of pain and symptom burden on the health-related quality of life of hemodialysis patients. J Pain Symptom Manage. 2010 Mar;39(3):477-85. doi: 10.1016/j.jpainsymman.2009.08.008. PMID 20303025
- [Background] Davison SN, Jhangri GS. The impact of chronic pain on depression, sleep, and the desire to withdraw from dialysis in hemodialysis patients. J Pain Symptom Manage. 2005 Nov;30(5):465-73. doi: 10.1016/j.jpainsymman.2005.05.013. PMID 16310620
- [Background] Murtagh FE, Addington-Hall J, Higginson IJ. The prevalence of symptoms in end-stage renal disease: a systematic review. Adv Chronic Kidney Dis. 2007 Jan;14(1):82-99. doi: 10.1053/j.ackd.2006.10.001. PMID 17200048
- [Background] Tong A, Crowe S, Chando S, Cass A, Chadban SJ, Chapman JR, Gallagher M, Hawley CM, Hill S, Howard K, Johnson DW, Kerr PG, McKenzie A, Parker D, Perkovic V, Polkinghorne KR, Pollock C, Strippoli GF, Tugwell P, Walker RG, Webster AC, Wong G, Craig JC. Research Priorities in CKD: Report of a National Workshop Conducted in Australia. Am J Kidney Dis. 2015 Aug;66(2):212-22. doi: 10.1053/j.ajkd.2015.02.341. Epub 2015 May 2. PMID 25943716
- [Background] Valderas JM, Kotzeva A, Espallargues M, Guyatt G, Ferrans CE, Halyard MY, Revicki DA, Symonds T, Parada A, Alonso J. The impact of measuring patient-reported outcomes in clinical practice: a systematic review of the literature. Qual Life Res. 2008 Mar;17(2):179-93. doi: 10.1007/s11136-007-9295-0. Epub 2008 Jan 4. PMID 18175207
- [Background] Basch E, Deal AM, Dueck AC, Scher HI, Kris MG, Hudis C, Schrag D. Overall Survival Results of a Trial Assessing Patient-Reported Outcomes for Symptom Monitoring During Routine Cancer Treatment. JAMA. 2017 Jul 11;318(2):197-198. doi: 10.1001/jama.2017.7156. PMID 28586821
- [Background] Denis F, Basch E, Septans AL, Bennouna J, Urban T, Dueck AC, Letellier C. Two-Year Survival Comparing Web-Based Symptom Monitoring vs Routine Surveillance Following Treatment for Lung Cancer. JAMA. 2019 Jan 22;321(3):306-307. doi: 10.1001/jama.2018.18085. PMID 30667494
- [Background] Naylor KL, Kim SJ, McArthur E, Garg AX, McCallum MK, Knoll GA. Mortality in Incident Maintenance Dialysis Patients Versus Incident Solid Organ Cancer Patients: A Population-Based Cohort. Am J Kidney Dis. 2019 Jun;73(6):765-776. doi: 10.1053/j.ajkd.2018.12.011. Epub 2019 Feb 6. PMID 30738630
- [Background] Weisbord SD, Fried LF, Mor MK, Resnick AL, Unruh ML, Palevsky PM, Levenson DJ, Cooksey SH, Fine MJ, Kimmel PL, Arnold RM. Renal provider recognition of symptoms in patients on maintenance hemodialysis. Clin J Am Soc Nephrol. 2007 Sep;2(5):960-7. doi: 10.2215/CJN.00990207. Epub 2007 Aug 8. PMID 17702730
- See also: Guidance for industry: patient-reported outcome measures: use in medical product development to support labeling claims: draft guidance — https://pubmed.ncbi.nlm.nih.gov/17034633/
- See also: Developing a Set of Core Outcomes for Trials in Hemodialysis: An International Delphi Survey — https://pubmed.ncbi.nlm.nih.gov/28238554/
- See also: Scope and Consistency of Outcomes Reported in Randomized Trials Conducted in Adults Receiving Hemodialysis: A Systematic Review — https://pubmed.ncbi.nlm.nih.gov/29475768/
- See also: Impact of pain and symptom burden on the health-related quality of life of hemodialysis patients — https://pubmed.ncbi.nlm.nih.gov/20303025/
- See also: The impact of chronic pain on depression, sleep, and the desire to withdraw from dialysis in hemodialysis patients — https://pubmed.ncbi.nlm.nih.gov/16310620/
- See also: The prevalence of symptoms in end-stage renal disease: a systematic review — https://pubmed.ncbi.nlm.nih.gov/17200048/
- See also: Research Priorities in CKD: Report of a National Workshop Conducted in Australia — https://pubmed.ncbi.nlm.nih.gov/25943716/
- See also: The impact of measuring patient-reported outcomes in clinical practice: a systematic review of the literature — https://pubmed.ncbi.nlm.nih.gov/18175207/
- See also: Overall Survival Results of a Trial Assessing Patient-Reported Outcomes for Symptom Monitoring During Routine Cancer Treatment — https://pubmed.ncbi.nlm.nih.gov/28586821/
- See also: Two-Year Survival Comparing Web-Based Symptom Monitoring vs Routine Surveillance Following Treatment for Lung Cancer — https://pubmed.ncbi.nlm.nih.gov/30667494/
- See also: Mortality in Incident Maintenance Dialysis Patients Versus Incident Solid Organ Cancer Patients: A Population-Based Cohort — https://pubmed.ncbi.nlm.nih.gov/30738630/
- See also: Renal provider recognition of symptoms in patients on maintenance hemodialysis — https://pubmed.ncbi.nlm.nih.gov/17702730/